CLINICAL TRIAL: NCT02259140
Title: ORCHID: Osteotomy vs Resection in CP Hip for Irreducible Dislocations: A Randomized Controlled Trial Comparing McHale to Castle Techniques
Brief Title: A Randomized Control Trial of Hip Dislocation Techniques for Pediatric Patients With Cerebral Palsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients have been enrolled since 2015. There has been difficulty recruiting patients for randomization. We have initiated a prospective cohort study evaluating salvage hip procedures for patients with cerebral palsy.
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Phoenix Children's Hospital (Other); The Hospital for Sick Children (Other); Boston Children's Hospital (Other); Children's Hospital of Michigan (Other); British Columbia Children's Hospital (Other); Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-199
Record Dates: First submitted 2014-07-14; First posted 2014-10-08 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Hip Dysplasia; Cerebral Palsy
Keywords: cerebral palsy; randomized controlled trial; hip dislocation; hip subluxation; patient centered outcomes; cost effectiveness analysis
MeSH Terms: conditions — Hip Dislocation; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proximal Femoral Resection Arthroplasty (Active Comparator): A 10-12 cm direct lateral incision will be made distally from the greater trochanter. The abductors of the hip are detached with sharp dissection. A capsulotomy is performed. The femur is exposed in a supra-periosteal manner (2 cm distal to the lesser trochanter) at the level of the ischium; transverse osteotomy will then be performed. The joint capsule will be sutured to itself. The iliopsoas tendon and the abductor tendons are attached to the capsule. The quadriceps will be brought around the proximal femoral stump and sutured to medial tissues.
  Interventions: Procedure: Proximal Femoral Resection Arthroplasty
- Subtrochanteric Valgus Osteotomy (Experimental): A 10-12 cm direct lateral incision will be made distally from the greater trochanter. The medial half of the abductors may be incised off the greater trochanter for repair. The femoral head is resected at the base of the neck. The ligamentum teres is incised off the head and preserved. A lateral closing wedge osteotomy is performed below the lesser trochanter. 3.5 or 4.5 5 hole locking/non-locking surgeon-contoured plate ( 45⁰) will be used to stabilize the osteotomy. Femoral torsion will be corrected. The psoas tendon will attach the ligamentum teres to the lesser trochanter. The anterior and posterior capsule is sutured together creating interposition tissue. If the ligamentum teres was sutured to the lesser trochanter, the capsule will not close, but will be covered by the psoas tendon.
  Interventions: Procedure: Subtrochanteric Valgus Osteotomy

INTERVENTIONS:
Procedure: Proximal Femoral Resection Arthroplasty — Drains will be placed at the surgeon's discretion. Patients will be placed in skin traction on the operative side. Post-operative bracing or casting will be at the surgeon's discretion. All patients will receive standardized post-operative prophylactic radiation to minimize heterotopic ossification.
  Other Names: Castle Technique
  Arms: Proximal Femoral Resection Arthroplasty
Procedure: Subtrochanteric Valgus Osteotomy — Drains will be placed at the surgeon's discretion. Post-operative bracing or casting will be at the surgeon's discretion. All patients will receive standardized post-operative prophylactic radiation to minimize heterotopic ossification.
  Other Names: McHale Technique
  Arms: Subtrochanteric Valgus Osteotomy

SUMMARY:
This randomized controlled trial will compare proximal femoral resection-interposition arthroplasty to proximal femoral resection with subtrochanteric valgus osteotomy for the treatment of painful irreducible hip dislocation in patients with cerebral palsy. The primary outcome is quality of life and care giver burden measured by The Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD) score at one year. Secondary outcomes will include pain (NCCPC-R, PROMIS pain intensity and PROMIS pain interference), function (mobility questions), complications and surgical parameters such as OR time and fluoroscopy time. A cost-effectiveness analysis will follow completion of the randomized controlled trial (RCT). The authors hypothesize that mean CPCHILD scores (measured at 1 year) will be significantly higher following the Subtrochanteric Valgus Osteotomy technique compared to Proximal Femoral Resection-Interposition Arthroplasty technique. Furthermore, the Proximal Femoral Resection-Interposition Arthroplasty technique will have a shorter length of hospital stay, shorter fluoroscopy and OR times and the Subtrochanteric Valgus Osteotomy will have longer sitting tolerance, less pain, smaller burden for caregivers, better health, and higher quality of life. Additionally the authors hypothesize that Subtrochanteric Valgus Osteotomy will be more expensive than Proximal Femoral Resection-Interposition Arthroplasty, due to the cost of the plate, longer operative time, longer length of stay, and blood loss, but Subtrochanteric Valgus Osteotomy will be preferred by patients due to less pain and better functional and quality of life outcomes.The results of this study are expected to improve outcomes for children with cerebral palsy with painful irreducible dislocated hips.

DETAILED DESCRIPTION:
The treatment of children with cerebral palsy (CP) with painful dislocated hips is a clinical challenge for the pediatric orthopedic surgeon. Although current regimens are based primarily on hip surveillance and early treatment of subluxation to avoid progression to dislocation, hip dislocations are still identified in the CP population. In younger children, in whom the hip is still of relatively normal morphology with intact cartilage and potential for remodeling (often identified by open tri-radiate cartilage) open hip reduction, varus rotational osteotomy and pelvic osteotomy may be a reasonable option. In older children, those with a deformed or damaged femoral head, those with closed triradiate cartilage, or in those with an irreducible hip, salvage options must be considered.

Multiple techniques exist for treatment of irreducible painful hips in CP, including proximal femoral resection-interposition arthroplasty, resection at the femoral neck with subtrochanteric valgus osteotomy, hip replacement or hip arthrodesis (fusing the femur to the socket in a static position). This wide variation in practices is consistent with clinical uncertainty regarding the optimal treatment method for this problem. The most frequently performed intervention for a painful irreducible hip in the setting of CP is a form of resection arthroplasty, either alone (proximal femoral resection-interposition arthroplasty) or in conjunction with valgus support osteotomy. Technique selection is based on the functional level of the patient, patient symptoms, and surgeon preference.{{257 Van Riet,A. 2009; 253 Wright,P.B. 2013}}

Although outcomes of resection at the femoral neck with subtrochanteric valgus osteotomy and proximal femoral resection-interposition arthroplasty techniques exist, published reports are retrospective non-randomized small series, which may be at risk for selection bias, and do not adequately capture all of the outcomes of interest, depending on what data has been routinely collected and documented in the medical chart.{{253 Wright,P.B. 2013; 259 Leet,A.I. 2005}},{{252 Boldingh,E.J. 2013}} Furthermore, results from these studies may be influenced by confounding factors, such as differences in patient age and other inequalities between groups at the time of surgery.{{252 Boldingh,E.J. 2013; 253 Wright,P.B. 2013; 277 Settecerri,J.J. 2000}} To the investigators knowledge, no prospective randomized comparison of hip resection techniques has been published accurately assessing child and parent quality of life, hip migration, or taking into account sitting and standing tolerance, pain, or hospital length of stay. Operative measures such as surgical time, blood loss and radiation exposure from intra-operative fluoroscopy have not previously been compared in a prospective manner.

This study was designed as a multicenter randomized trial to answer an important clinical question about a rare condition, and to do so with a clearly defined objective and validated set of outcomes. This simple trial can be executed on a relatively small budget with simple outcome measures, and recruitment of a small number of patients at each of a few centers well equipped for research. By involving multiple surgeons and patients from various geographies, we improve the generalizability of this study. Our institution and collaborating institutions have been successful in completing randomized clinical trials in the past. This study will answer a clinical question that is important and current, providing orthopedic surgeons with an evidence-based answer: the optimal technique in treating painful irreducible hip dislocation in patients with cerebral palsy. The proposed research study aims to fill these gaps.

ELIGIBILITY:
Inclusion Criteria:

* 7-21 years of age
* Painful irreducible Hip dislocation and cerebral palsy diagnosis
* GMFCS 4 or 5

Exclusion Criteria:

* GMFCS 1-3
* Decline to participate
* Outcome scales not validated in patient language.
* Candidate for total hip replacement

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2020-09 (Estimated); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life and Caregiver Burden | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Measured by CPCHILD.

SECONDARY OUTCOMES:
Mean Hip Migration | Baseline, post-operative, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  X-rays measuring hip migration will be standardized to anteroposterior (AP) Pelvis and Frog lateral. Patient positioning will be standardized according to normal clinical practice.
Pain Scores | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  NCCPC-R, PROMIS Pediatric Pain Interference, PROMIS Pediatric Pain Intensity
Caregiver Burden | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Indirect Cost Form
Length of Stay | An expected average of 5 days
  Discharge date - admission date. Transform into number of days. Length of stay can vary from days to weeks, if serious complication occurs.
Sitting Tolerance | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Measured by wheelchair pressure mapping (hours /wk)
Range of Motion | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Measured by goniometer (degrees)
Complications | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Infection, deep vein thrombosis (DVT), fracture, heterotropic calcification
Function | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Measured by GMFCS.
Splint | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Need for splint or cast will be documented in medical records.
Secondary Surgery | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Need for secondary surgery will be documented in medical records.
Standing Tolerance | Baseline, 2-6 weeks, 5-7 months, 11-13 months and 23-25 months
  Measured by instander (hours/ week)
Medical Costs | 4 years (end of study)
  analyze claims data (approx 4 years)
Operative Outcomes | intra-operative
  radiation, total time during surgery, skin dose, blood loss, surgeon experience, hip resection technique

CONTACTS AND LOCATIONS:
Overall Officials: Emily Dodwell, MD MPH FRCSC, Principal Investigator — Hospital for Special Surgery, New York
Locations (7):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Miami Children's Hospital, Miami, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Hospital for Special Surgery, New York, New York
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Background] Van Riet A, Moens P. The McHale procedure in the treatment of the painful chronically dislocated hip in adolescents and adults with cerebral palsy. Acta Orthop Belg. 2009 Apr;75(2):181-8. PMID 19492557
- [Background] Wright PB, Ruder J, Birnbaum MA, Phillips JH, Herrera-Soto JA, Knapp DR. Outcomes after salvage procedures for the painful dislocated hip in cerebral palsy. J Pediatr Orthop. 2013 Jul-Aug;33(5):505-10. doi: 10.1097/BPO.0b013e3182924677. PMID 23752147
- [Background] Leet AI, Chhor K, Launay F, Kier-York J, Sponseller PD. Femoral head resection for painful hip subluxation in cerebral palsy: Is valgus osteotomy in conjunction with femoral head resection preferable to proximal femoral head resection and traction? J Pediatr Orthop. 2005 Jan-Feb;25(1):70-3. doi: 10.1097/00004694-200501000-00016. PMID 15614063
- [Background] Boldingh EJ, Bouwhuis CB, van der Heijden-Maessen HC, Bos CF, Lankhorst GJ. Palliative hip surgery in severe cerebral palsy: a systematic review. J Pediatr Orthop B. 2014 Jan;23(1):86-92. doi: 10.1097/BPB.0b013e3283651a5d. PMID 24025529
- [Background] Settecerri JJ, Karol LA. Effectiveness of femoral varus osteotomy in patients with cerebral palsy. J Pediatr Orthop. 2000 Nov-Dec;20(6):776-80. doi: 10.1097/00004694-200011000-00015. PMID 11097253